CLINICAL TRIAL: NCT04341402
Title: Dr. Bill Antifungal Nail Gel Study
Brief Title: Systemic Uptake of Diclofenac Sodium in Combination With Miconazole as Antifungal Nail Gel When Applied Daily With Monitoring of Hepatic and Renal Enzymes, and Serum Levels of Diclofenac 12 Hours After Application, and at 3 and 6 Months Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: William N Handelman (Other)
Responsible Party: Sponsor-Investigator, William N Handelman, Principal Investigator, Bay Area Medical
Organization: Bay Area Medical (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IORG0010258
Record Dates: First submitted 2020-02-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Tinea Unguium, Onychomycosis
Keywords: Toenail fungus
MeSH Terms: conditions — Onychomycosis | interventions — Diclofenac; Miconazole; Urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): miconazole 3% & diclofenac sodium 1% & urea 40% in topical gel daily for 6 months.
  Interventions: Drug: Antifungal Nail Gel Study

INTERVENTIONS:
Drug: Antifungal Nail Gel Study — Daily Application antifungal gel of miconazole 3% and diclofenac sodium 1% and urea 40% to infected nails.
  Other Names: drug: diclofenac sodium; drug: miconazole; drug: urea

SUMMARY:
Study evaluates these take of diclofenac sodium when used in conjunction with miconazole and urea as a topical antifungal nail gel treatment for onychomycosis. All of the patient's will be treated with the active formula and blood levels of diclofenac sodium tested for as well as monitoring of hepatic and renal functions

DETAILED DESCRIPTION:
Tinea Unguium/onychomycosis is a ubiquitous health problem affecting ~3% of the adult population. It is associated with higher risk for other disease processes. Effective treatment for this disease has been lacking. Oral antifungal agents are associated with high incidence of recurrence of disease, hepatotoxicity, cytochrome P450 Pathway interference, non-compliance, side effects and cost. No effective long-term topical applications have been verified. Debridement of the damaged nail in combination with a broad-spectrum topical antifungal agent and an anti-inflammatory agent is a safe, inexpensive and easily formulated alternative to previous ineffective treatments. The rationale for debridement is simple in that the effectiveness of the topical antifungal is present only when it is in contact with the fungal agent, nail bed and involved diseased tissue. The associated inflammatory response associated with fungal infections is well-established. The only topical NSAID available in the United States is diclofenac sodium. The combination of miconazole, diclofenac sodium and urea has proven effective in this researcher's self-treatment of tinea unguium. Miconazole and diclofenac sodium are well studied and well-established pharmaceutical

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 21 years of age at Visit 1.
2. Not pregnant.
3. Stage 3 or lower Chronic Renal Failure.
4. PT/INR < 1.3 and not on anti-thrombotic; AST, ALT, Total Bilirubin WNL.
5. Documentation of a diagnosis of tinea unguium as evidenced by one or more clinical features consistent with the onychomycosis and one or more of the following criteria: KOH prep of the nail scrapings or positive culture of the nail scrapings; culture of nail with growth of any of the following Dermatophytes, non-dermatophytes or yeast.
6. TABLE 1 Epidermophyton floccosum Trichophyton mentagrophytes Trichophyton rubrum Acremonium Alternaria species Aspergillus species Botryodiplodia theobromae Fusarium species Onycochola canadensis Pyrenochaeta unguis-hominis Scytalidium dimidiatum scopulariopsis species Scytalidium hyalimum Candida albicans

Exclusion Criteria:

1. Chronic renal failure, chronic liver disease, alcoholism, pregnant, breastfeeding, or unwilling to practice birth control during participation in the study if of childbearing age..
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Concomitant use of any prescribed medication that may be adversely affected by diclofenac sodium.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Diclofenac sodium serum levels | 12 hours
  Peak Plasma Concentration (Cmax) diclofenac sodium 12 hours after 1st dose

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of diclofenac sodium 3 months after starting application | 3 months
  Peak Plasma Concentration (Cmax) of diclofenac sodium

CONTACTS AND LOCATIONS:
Overall Officials: William N Handelman, MD, Principal Investigator — Bay Area Medical
Locations (1):
- Bay Area Medical, St. Petersburg, Florida, United States